CLINICAL TRIAL: NCT03404986
Title: Ultrasound Guided Ureteroscopy for the Treatment of Lower Third Ureteric Stones in Adults
Brief Title: Ultrasound Guided Ureteroscopy and Ureteric Stones
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohamed Loay, Resident, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: USUUS
Record Dates: First submitted 2018-01-14; First posted 2018-01-19 (Actual); Last update posted 2022-12-05 (Actual); Status verified 2022-12

CONDITIONS: Ureteric Stone
MeSH Terms: conditions — Ureterolithiasis | interventions — Ureteroscopy; High-Energy Shock Waves

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standardized ureteroscopy group (Other)
  Interventions: Procedure: ureteroscopy
- Ultrasonography ureteroscopy group (Other)
  Interventions: Procedure: ureteroscopy; Radiation: Ultrasonography

INTERVENTIONS:
Procedure: ureteroscopy — The patients will be subjected to rigid ureteroscopy
Radiation: Ultrasonography — The patients will be subjected to Ultrasonography
  Arms: Ultrasonography ureteroscopy group

SUMMARY:
The prevalence of urolithiasis is steadily increasing with an estimation of 1 out of 11 people in the United States. The prevalence of calculi in Afro-Asian region including Arab Republic of Egypt ranges from 4% to 20%. Ureteroscopy is one of the first line treatments for definitive management of ureteric stones. Conventional ureteroscopy relies on intraoperative fluoroscopy for visualization and guidance, exposing the patient, surgeon and operating room staff to ionizing radiation. To minimize the hazards of ionizing radiation there has been a trend toward radiation free alternative imaging modalities . Ultrasound provides an excellent alternative for upper urinary tract imaging because it is radiation free, rapid, portable and allows excellent visualization of the renal pelvis and calyces. There is increasing awareness and concern about the clinical use of ionizing radiation and the need to decrease exposure of patients and medical professionals. Ultrasound guided ureteroscopy in pregnant females and children- in whom fluoroscopy is to be minimized or avoided when possible - has been reported.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with single symptomatic lower third ureteric radio-opaque stones indicated for endoscopic treatment.
2. Age group 18 years old or above.
3. Stone size 15 mm or less.

Exclusion Criteria:

1. Patients with bilateral ureteric stones
2. Ureteric congenital anomalies e.g. double ureter and ectopic ureter.
3. Previously failed ureteroscopy or previous ureteroneocystostomy.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2020-04-01 (Actual); Study Completion 2020-04-01 (Actual)

PRIMARY OUTCOMES:
Number of patients treated effectively by the two methods | 1 hour

CONTACTS AND LOCATIONS:
Locations (1):
- Women Health Hospital - Assiut university, Asyut, Egypt